CLINICAL TRIAL: NCT00817453
Title: Cross-Sectional Cohort Study of Laboratory and Clinical Patterns in Early PD
Brief Title: Early Parkinson's Disease (PD) Cross-Sectional
Acronym: EPDX
Status: Terminated | Type: Observational
Why Stopped: All subjects transferred to long term study NCT00817726 RBD Longitudinal
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Mya Schiess, MD, The University of Texas Health Science Center, Houston
Other Study IDs: SchiessEPDX2008
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — CSF and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Clinically diagnosed Early iPD
- 2: Age/gender matched controls without neurodegenerative diagnosis
- atypical or late Parkinsonian Syndromes: Includes subjects facing or having undergone DBS, diagnoses of MSA, PSP or other atypical syndromes.

SUMMARY:
Purpose:

1. To see if cytokine levels and oligomeric alpha-synuclein levels in blood and cerebrospinal fluid could be used as biological markers for Parkinson's disease (PD) onset and progression.
2. To characterize and define patterns in the clinical features of sleep, olfactory function and motor function in the early stages of idiopathic (sporadic) Parkinson's disease (PD)and atypical or late Parkinsonian Syndromes.

Procedures:

All subjects, control,early PD diagnosis and atypical or late Parkinsonian Syndromes, will have 1) a medical and neuro history and physical including videotaping of movements, 2) neuropsychological testing, 3) a sleep study, 4) olfactory (sense of smell) testing, 5)blood draw and LP for serum and CSF testing, & 6) functional MRI. All of these procedures are often done in the diagnosis of PD. Any test performed prior to enrollment as part of the clinical evaluation may be used in place of repeating the procedure. Subjects will have 1 set of study visits (up to 3 visits) in order to accomplish a complete set of data.

ELIGIBILITY:
Inclusion Criteria:

1. 35-80 year old men & women
2. Patients with iPD or Parkinsonian syndromes, or controls consisting of healthy subjects, or subjects who have a non-neurodegenerative diagnosis but are otherwise healthy.
3. Gives written informed consent
4. Pregnant women are not excluded, but will be identified by HCG.

Exclusion Criteria:

1. Parkinsonian symptoms not due to idiopathic (sporadic) PD, such as those that are medication induced, toxic substance induced or representative of an atypical Parkinsonian syndrome will be categorized separately.
2. Any unstable or uncontrolled medical or psychiatric condition.
3. Renal (creatinine over 1.6) or hepatic insufficiency (LFT three-fold higher than normal range), or a history of significant cardiac disease.
4. If there is a history or evidence of coagulopathy, on medications such as Plavix, Aggrenox, heparin, coumadin, or large doses of aspirin, must be able to remain off these medications for at least 3 days, and have stable blood coagulation values prior to any lumbar puncture (LP).
5. Significant dementia (MMSE<25/30 or MOCA<25/30) that would interfere with study procedures or the giving of informed consent for the study .
6. Active infections including skin, respiratory or GI infections, and HIV+ (if undergoing an LP).
7. Any evidence of a different neurodegenerative disorder, for example, Alzheimer's Disease or Huntington's Disease.
8. fMRI will not be performed is screening questionnaire identifies a reason.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: clinical diagnosis of early PD and age/gender matched controls
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
1) Quantify and compare levels of IL-6, 2, 4,10 and IL-1 beta,IFN,TNF alpha, soluble monomeric alpha-synuclein and oligomeric alpha-synuclein in the CSF and serum of the early PD patients compared to age- and sex-matched controls. | 2 years
2) Characterize the sleep, olfactory,medical and neurologic assessments of early symptomatic PD subjects compared to age- and sex-matched normal controls. | 2 years

SECONDARY OUTCOMES:
Ability of functional MRI to show distinct features for PD | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mya C Schiess, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] Schiess M, Oh I. Serum uric acid and clinical progression in Parkinson disease: potential biomarker for nigrostriatal failure. Arch Neurol. 2008 Jun;65(6):698-9. doi: 10.1001/archneur.65.6.698. No abstract available. PMID 18541788
- [Background] Bick RJ, Poindexter BJ, Kott MM, Liang YA, Dinh K, Kaur B, Bick DL, Doursout MF, Schiess MC. Cytokines disrupt intracellular patterns of Parkinson's disease-associated proteins alpha-synuclein, tau and ubiquitin in cultured glial cells. Brain Res. 2008 Jun 27;1217:203-12. doi: 10.1016/j.brainres.2008.03.081. Epub 2008 Apr 10. PMID 18501880
- [Background] Hood AJ, Amador SC, Cain AE, Briand KA, Al-Refai AH, Schiess MC, Sereno AB. Levodopa slows prosaccades and improves antisaccades: an eye movement study in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2007 Jun;78(6):565-70. doi: 10.1136/jnnp.2006.099754. Epub 2006 Dec 18. PMID 17178817
- [Background] Schiess M. Nonsteroidal anti-inflammatory drugs protect against Parkinson neurodegeneration: can an NSAID a day keep Parkinson disease away? Arch Neurol. 2003 Aug;60(8):1043-4. doi: 10.1001/archneur.60.8.1043. No abstract available. PMID 12925357
- [Background] Schiess MC, Zheng H, Soukup VM, Bonnen JG, Nauta HJ. Parkinson's disease subtypes: clinical classification and ventricular cerebrospinal fluid analysis. Parkinsonism Relat Disord. 2000 Apr 1;6(2):69-76. doi: 10.1016/s1353-8020(99)00051-6. PMID 10699387